CLINICAL TRIAL: NCT01461850
Title: Surgical Complications Related to Primary or Interval Debulking in Ovarian Neoplasm
Acronym: SCORPION
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Prof. Giovanni Scambia, Professor, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 789/11
Record Dates: First submitted 2011-10-19; First posted 2011-10-28 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Stage IIIC Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Neoadjuvant Therapy; Chemotherapy, Adjuvant

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned (1:1 ratio) to undergo either PDS followed by systemic adjuvant chemotherapy, or NACT followed by IDS. Random assignment will be centralised at the Institutional clinical trial center using a block-randomisation computer-generated list (maximum allowable percentage deviation = 10%). Allocation will be concealed to patients and investigators. Patients and investigators will not be masked to group assignment.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Primary debulking surgery (Active Comparator): All patients with suspicion of advanced ovarian carcinoma (FIGO stage IIIC) will undergo to a diagnostic laparoscopy in order to obtain a laparoscopic score (PIV) based on seven parameters: omental cake, peritoneal and diaphragmatic extensive carcinosis, mesenteric retraction, bowel and stomach infiltration, spleen and/or liver superficial metastasis, as previously published (Fagotti et al, American Journal of Obstetrics and Gynecology, 2008) Patients with PIV ≥ 8 and ≤ 12 randomized in this group will be submitted to an attempt of primary debulking surgery in order to obtain RT < 1 cm, followed by adjuvant chemotherapy.
  Interventions: Procedure: Primary Debulking Surgery + Adjuvant Chemotherapy
- Interval debulking surgery (Experimental): All patients with suspicion of advanced ovarian carcinoma (FIGO stage IIIC) will undergo to a diagnostic laparoscopy in order to obtain a laparoscopic score (PIV) based on seven parameters: omental cake, peritoneal and diaphragmatic extensive carcinosis, mesenteric retraction, bowel and stomach infiltration, spleen and/or liver superficial metastasis, as previously published (Fagotti et al, American Journal of Obstetrics and Gynecology, 2008) Patients with PIV ≥ 8 and ≤ 12 randomized in this group will be submitted only to diagnostic laparoscopy followed by neoadjuvant chemotherapy and subsequent Interval Debulking Surgery, followed by further cycles of chemotherapy.
  Interventions: Drug: Neoadjuvant chemotherapy + Interval Debulking Surgery

INTERVENTIONS:
Drug: Neoadjuvant chemotherapy + Interval Debulking Surgery — Patients with suspected advanced ovarian cancer (FIGO stage IIIC) will undergo only to diagnostic laparoscopy. Omental cake, diaphragmatic or peritoneal extensive carcinomatosis, tumor diffusion to the small and large curvature of the stomach, large and/or small bowel mesentery disease, spleen and/or liver metastases will be investigated in order to obtain a laparoscopic score. After neoadjuvant chemotherapy interval debulking surgery will be performed: total hysterectomy, bilateral salpingo-oophorectomy, radical omentectomy, appendectomy, pelvic and paraaortic lymphadenectomy, eventual bowel resection, eventual bladder resection, eventual splenectomy, eventual parietal and diaphragmatic peritonectomy, eventual gastric resection, eventual hepatic resection, eventual pancreas resection, eventual cholecystectomy.
  Arms: Interval debulking surgery
Procedure: Primary Debulking Surgery + Adjuvant Chemotherapy — Patients with suspected advanced ovarian cancer (FIGO stage IIIC) will undergo to diagnostic laparoscopy. Omental cake, diaphragmatic or peritoneal extensive carcinomatosis, tumor diffusion to the small and large curvature of the stomach, large and/or small bowel mesentery disease, spleen and/or liver metastases will be investigated in order to obtain a laparoscopic score. Then, an attempt of laparotomic cytoreduction will be performed: total hysterectomy, bilateral salpingo-oophorectomy, radical omentectomy, appendectomy, pelvic and paraaortic lymphadenectomy, eventual bowel resection, eventual bladder resection, eventual splenectomy, eventual parietal and diaphragmatic peritonectomy, eventual gastric resection, eventual hepatic resection, eventual pancreas resection, eventual cholecystectomy.
  Arms: Primary debulking surgery

SUMMARY:
Patients with advanced ovarian cancer (FIGO stage III C) and highly disseminated tumor will be randomized into two arms: primary debulking surgery followed by adjuvant chemotherapy vs. neoadjuvant chemotherapy followed by interval debulking surgery (IDS). The primary end point is the evaluation and comparison of the surgical complications of primary surgery and IDS and the evaluation of the progression free survival (PFS)

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected advanced ovarian cancer (FIGO stage IIIC)
* PIV ≥ 8, PIV ≤ 12
* Estimated life expectancy of at least 4 weeks.
* PS ≤ 2
* Appropriate respiratory, hepatic, cardiological, bone marrow and renal functions (Creatinine Clearance > 60 mL/min according to Cockcroft formula)
* Patient capable of consent.

Exclusion Criteria:

* Pregnancy or breastfeeding.
* Non-appropriate respiratory, hepatic, cardiological, bone marrow and renal functions
* Large size mass reaching the xiphoid, occupying all the abdominal cavity and/or infiltrating the abdominal wall.
* Mesenteric retraction

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2011-10-01 (Actual); Primary Completion 2014-11-30 (Actual); Study Completion 2016-05-31 (Actual)

PRIMARY OUTCOMES:
Evaluation and comparison of early surgical complications of primary surgery and Interval debulking surgery. | thirty days
  Early surgical complications:
  * Blood transfusion
  * Re-laparotomy
  * suture dehiscence of laparotomy.
  * Venous thrombosis
  * Haemorrhage
  * Death in the post-operative period
  * Digestive fistula
  * Urinary fistula
  * Lymphocyst
  * Fever
  * Infection
  * Pleural effusion
  * Pulmonary embolism
  * Pneumothorax
  * Pneumonia
Evaluation and comparison of late surgical complications of primary surgery and Interval debulking surgery | six months
  Late surgical complication:
  * Death for every reason.
  * Suture dehiscence of laparotomy with opening of the abdominal muscles
  * Fever due to lymphocystis infection
Evaluation of the progression free survival (PFS) | Thirty-six months
  Time from randomization until recurrence of tumor or death from any cause.

SECONDARY OUTCOMES:
Overall Survival | Thirty-six months
  Time from randomization until death from any cause.
Evaluation of Quality of life | 12 months
  Quality of life will be assess using the EORTC quality of life questionnaire core-36 (QLQC-30) and the ovarian cancer-specific quality of life questionnaire (QLQ-Ov28). These will be complete at study entry, at the 4th cycle or before IDS (in arm A and arm B, respectively), at the 6th cycle, and 6 months after the last cycle of chemotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of the Sacred Heart, Rome, Italy

REFERENCES:
- [Result] Vergote I, Trope CG, Amant F, Kristensen GB, Ehlen T, Johnson N, Verheijen RH, van der Burg ME, Lacave AJ, Panici PB, Kenter GG, Casado A, Mendiola C, Coens C, Verleye L, Stuart GC, Pecorelli S, Reed NS; European Organization for Research and Treatment of Cancer-Gynaecological Cancer Group; NCIC Clinical Trials Group. Neoadjuvant chemotherapy or primary surgery in stage IIIC or IV ovarian cancer. N Engl J Med. 2010 Sep 2;363(10):943-53. doi: 10.1056/NEJMoa0908806. PMID 20818904
- [Result] Fagotti A, Ferrandina G, Fanfani F, Garganese G, Vizzielli G, Carone V, Salerno MG, Scambia G. Prospective validation of a laparoscopic predictive model for optimal cytoreduction in advanced ovarian carcinoma. Am J Obstet Gynecol. 2008 Dec;199(6):642.e1-6. doi: 10.1016/j.ajog.2008.06.052. Epub 2008 Sep 17. PMID 18801470
- [Result] Fagotti A, Ferrandina G, Fanfani F, Ercoli A, Lorusso D, Rossi M, Scambia G. A laparoscopy-based score to predict surgical outcome in patients with advanced ovarian carcinoma: a pilot study. Ann Surg Oncol. 2006 Aug;13(8):1156-61. doi: 10.1245/ASO.2006.08.021. Epub 2006 Jun 21. PMID 16791447
- [Derived] Fagotti A, Ferrandina MG, Vizzielli G, Pasciuto T, Fanfani F, Gallotta V, Margariti PA, Chiantera V, Costantini B, Gueli Alletti S, Cosentino F, Scambia G. Randomized trial of primary debulking surgery versus neoadjuvant chemotherapy for advanced epithelial ovarian cancer (SCORPION-NCT01461850). Int J Gynecol Cancer. 2020 Nov;30(11):1657-1664. doi: 10.1136/ijgc-2020-001640. Epub 2020 Oct 7. PMID 33028623
- [Derived] Fagotti A, Vizzielli G, Fanfani F, Costantini B, Ferrandina G, Gallotta V, Gueli Alletti S, Tortorella L, Scambia G. Introduction of staging laparoscopy in the management of advanced epithelial ovarian, tubal and peritoneal cancer: impact on prognosis in a single institution experience. Gynecol Oncol. 2013 Nov;131(2):341-6. doi: 10.1016/j.ygyno.2013.08.005. Epub 2013 Aug 9. PMID 23938372